CLINICAL TRIAL: NCT04725578
Title: Evaluating the Telehealth Single Session Consultation Service
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2019-00362-2
Record Dates: First submitted 2021-01-18; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Mental Health Impairment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Single Session Consultation (Experimental)
  Interventions: Behavioral: Telehealth Single Session Consultation

INTERVENTIONS:
Behavioral: Telehealth Single Session Consultation — A remotely delivered, single, goal-directed consultation session based on Solution-Focused Brief Therapy (SFBT). SFBT is an evidence-based therapy approach that is primarily focused on the client's present problems and their immediate future. When using SFBT in a single-session the aim of the intervention becomes empowering the client to take the smallest possible steps towards their desired future.
  Other Names: Telehealth-SSC

SUMMARY:
Stony Brook University is home to several mental health clinics, that all work towards achieving overall wellness of their clients. The goals of Stony Brook University are met with the help of associated clinics that strive to improve wellness of individuals and their communities by helping to treat both mental and physical health impairments. One of these many clinics is the Krasner Psychological Center (KPC).

At present, the KPC faces a challenge common to virtually all mental health clinics across the United States: the demand for psychological services far outpaces the number of available providers. Indeed, in the US, approximately 70% of those in need of mental health services do not receive them. As such, wait-lists at mental health clinics like the KPC are increasingly long, and longer wait-times for psychotherapy have predicted worse clinical outcomes once treatment is accessed (i.e., a 'nocebo' effect). Thus, there is a pressing need for effective, sustainable service delivery models that may facilitate more rapid access to care-for instance, providing a low-intensity service rapidly after an individual decides to seek treatment, capitalizing on client motivation. This sort of rapidly-provided, low-intensity service might have the added benefit of reducing overall waitlist lengths--e.g., if some subset of clients find the low-intensity service to be sufficient, a single session might be sufficient (in some cases) to spur positive behavioral and emotional change.

One solution to this problem is the integration of single-session services into mental health clinics. Extensive research suggests that both youths and adults can benefit from just one session of goal-directed counseling, and these clinical benefits have been observed for a wide array of problems-including anxiety, depression, self-harm, and interpersonal conflicts. This research suggests the possibility that, for some subset of clients, a single session of counseling may be helpful, or even sufficient, in reducing clinical distress. Further, offering such service in a telehealth format will alleviate frequently cited barriers to care like transportation, geographic constraints, and limited time.

Therefore, the objective of this study is to examine the feasibility, acceptability, and short-term effects of the new telehealth-Single-Session Consultation (SSC) service, which is presently being provided to clients on the waiting list for psychotherapeutic services at the Krasner Psychological Center. The telehealth-SSC offers clients the opportunity to participate in a single, goal-directed consultation session based on Solution-Focused Brief Therapy (SFBT) within two weeks of inquiring about services at the KPC (typically, clients wait 2-6 months prior to their initial clinic appointment). SFBT is an evidence-based therapy approach that guides services offered by existing single-session therapy clinics internationally. Clients who participate in the telehealth-SSC at any of these clinics may find the session helpful; two weeks after participating in the session, they receive the option to remain on the waitlist for long-term psychotherapy or remove themselves from the waitlist for psychotherapy, depending on whether they feel their clinical needs have been successfully addressed.

DETAILED DESCRIPTION:
The Stony Brook University (SBU) clinical psychology doctoral program is currently ranked 4th among the top clinical psychology doctoral programs in the country (2016, U.S. News and World Report, Best Graduate Schools) and is accredited by both the APA Committee on Accreditation (APA CoA) and the Psychological Clinical Science Accreditation System (PCSAS). The Krasner Psychological Center (KPC) is a psychology training clinic housed in the Department of Psychology and associated with the doctoral program in clinical psychology at SBU. The mission of the KPC is twofold, namely, (a) to provide high quality experiential training in the delivery of psychological services to trainees in the associated 3 doctoral program, as well as to externs, doctoral interns, and post-doctoral residents; and (b) to provide evidence-based mental health services to the nearby communities. All supervisors at the KPC are doctoral-level psychologists. Psychotherapy services at the KPC are based on Cognitive-Behavior Therapy models and include weekly, outpatient psychotherapy for a wide range of problems in children and adults; therapy is designed to be short-term, personalized, and effective in empowering clients to manage their symptoms and distress.

The telehealth-single-session consultation, a one-time service provided to adolescents and adults (13+) on the clinics' waitlist (which may extend from 2 to 6 months), includes components of Solution-Focused Brief Therapy (SFBT). SFBT lends itself naturally to the single-session format in that it focuses on the present and future, targeting the desired outcome of therapy, a future in which the primary problem is absent or less influential. Importantly, SFBT providers focus on the factors that maintain/underlie solutions rather than the factors than maintain/underlie problems.

GENERAL SCREENING PROCEDURES

When individuals seeking services at the KPC express interest in scheduling an appointment with a clinician, they are first instructed (by phone) about the clinical and research aims by the clinic's staff. The clinical staff is a trained, independent member and is not involved in the provision of psychotherapy or single-session consultation services. The clinical staff conducts a standardized, structured phone screen with the individual to identify primary reasons for seeking mental health services and to assess the appropriateness of presenting concerns for treatment at the KPC. If the individual is eligible to receive services at the KPC (i.e., if their concerns fall within the scope of clinical problems treated; if the individual/family is English-speaking; and if problems are not so acute as to require immediate hospitalization, in which case they are referred to the nearest emergency room), the client is placed on the waitlist for psychotherapy services.

During the same phone call, if the identified patient is 13 years or older, the clinic staff then introduces the opportunity to participate in the telehealth-Single Session Consultation (SSC) service at the KPC.

The clinic staff indicates that as part of telehealth-SSC service participation the client will be asked to complete questionnaires in order to provide their clinician with information about their current mental health, and for the purposes of planning and assessing the usefulness of services. The clinic staff will also indicate that the individual may opt to allow or not allow us to use this data for research purposes. They will be informed that if they do choose to allow their data to be used for research, it will be de-identified and combined with other patient data for the purposes of understanding how well our treatment programs work for different types of individuals. The staff will emphasize that their choice to participate, or not participate in research will NOT impact their eligibility for the telehealth-SSC service or longer-term psychotherapy in any way.

The clinician will obtain fully informed consent via Qualtrics prior to the SSC appointment. Adult patients (or adolescent patient and her/his parent) can either agree or disagree to allow the research team to use their clinical data for research by checking the appropriate check-box on the consent form. Patients will also be able to elect to participate in the specific study described in the consent form and/or to have their de-identified data added to a registry for future unspecified research projects.

DATA COLLECTION PROCEDURES SPECIFIC TO THE TELEHEALTH-SINGLE-SESSION CONSULTATION SERVICE

Immediately prior to telehealth-SSC participants will be asked to complete the following via a Qualtrics survey:

* PHQ-9
* GAD-7
* Beck Hopelessness Scale - 4 item
* Readiness for Change Rulers

Immediately following the one-hour telehealth-SSC session, participants will be asked to complete the following via a Qualtrics survey:

* Consultation Feedback Form
* Working Alliance Inventory Short Form - client
* Beck Hopelessness Scale - 4 item
* Readiness for change Ruler

Finally, two weeks after completing the telehealth-SSC, participants will be followed-up with a Qualtrics survey containing:

* PHQ-9
* GAD-7

NOTE 1: A client may reschedule an SSC session if they are unable to attend it. The KPC will not limit the number of times a client is permitted to reschedule an SSC session, should they remain interested in receiving one. Additionally, if clients endorse significant clinical risk (to themselves or others) while participating in the study, study procedures may be interrupted (e.g., an SSC session may be terminated in order to address urgent clinical needs). If a client's initial SSC session is interrupted or terminated due to a need to address urgent clinical risk, the client will be permitted to reschedule their SSC session for a later date.

NOTE 2: If a participant does not respond to the clinic's requests for a 2-week follow-up within two weeks of being contacted, per KPC policy, it will be assumed that the client is no longer interested in services and will be removed from the waiting list. Pre-to-post SSC data for these clients will still be used for analyses unless they request that their data not be used in the study.

NOTE 3: The lead investigator (Jessica Schleider) will train all SSC clinicians prior to their delivering SSC sessions with clients. This training will be approximately 2 hours in length and will review the principles and key elements of the SSC protocol, in addition to challenges that might emerge while delivering the SSC.

ELIGIBILITY:
Inclusion Criteria:

* All adolescent (ages 13+) and adult clients on the waitlist for clinical psychotherapy services at the KPC will be eligible to take part in this research.

Exclusion Criteria:

* Child clients at the KPC under the age of 13 will not be eligible to participate in this study, because the teletherapy-Single-Session Consultation service presently being offered at the KPC is designed for use with adolescents and adults (i.e., it would be developmentally inappropriate for younger children.).
* Non-English speaking individuals will not be eligible to receive any clinical services at the KPC because all therapists at the clinics are English-speaking.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in PHQ-9 | Baseline & 2-week follow-up
  The PHQ-9 asks participants to rate 9 questions assessing dimensions of depression on a scale of 0 (Not at all) to 3 (Nearly every day). Total score ranges from 0 to 27 with higher scores indicating higher levels of depression.
Change in GAD-7 | Baseline & 2-week follow-up
  The GAD-7 asks participants to rate 7 statements based on how generally anxious they have felt over the past 2 weeks on a 4 point scale ranging from 0 (Not at all) to 3 (Nearly every day). Total score ranges from 0 to 21 with higher scores representing higher generalized anxiety.
Change in Beck Hopelessness Scale | Baseline & 2-week follow-up
  Respondents report agreement with 4 items, each rated on a 0 (Very False) to 3 (Very True) scale, indicating levels of hopelessness about the future. Higher summed scores reflect greater levels of hopelessness with total scores ranging from 0-12.
Change in Readiness for Change Ruler | Baseline & immediately Post-SSC
  The readiness for change ruler is a 3 item measure that examines participant's willingness to change to improve their mental health on a 0 (not at all confident/important/ready) to 10 scale (completely confident/ready). The total score ranges from 0 to 30, with higher score indicating higher levels of willingness to change.

SECONDARY OUTCOMES:
Working Alliance Inventory - Short | Immediately Post-SSC
  The working alliance inventory asks participants to rate 12 statements regarding their personal experiences they had with their therapist on a scale of 1 (Never) to 7 (Always). The overall score will be a single mean score (possible range: 1-7; items 4 and 10 are reversed scored) reflecting patient-rated working alliance with their therapist. Higher scores reflect a stronger perceived therapeutic alliance.
Consultation Feedback Form | Immediately Post-SSC
  The consultation feedback form contains 5 items, rated on a 1 ("Not at all") to 5 ("Very much") Likert scale, indicating endorsement of a series of statements about responses to the Single Session Consultation program (e.g., "Did you find the consultation helpful in addressing your concern(s)?" and "How hopeful are you that the action plan will be useful?"). Higher mean scores across these 5 items indicate greater perceived usefulness of the SSC.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available on Open Science Framework upon conclusion of the study
Supporting Information: Study Protocol, SAP, Analytic Code

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT04725578/SAP_000.pdf